CLINICAL TRIAL: NCT00396994
Title: Low Magnitude Mechanical Stimulation (LMMS) to Improve Bone Mineral Density (BMD)
Brief Title: "VIBES"--Low Magnitude Mechanical Stimulation to Improve Bone Mineral Density
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hebrew SeniorLife (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Douglas Kiel, Director Musculoskeletal Research Center, Hebrew SeniorLife
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: AG0071; R01AG025489 (NIH)
Record Dates: First submitted 2006-11-07; First posted 2006-11-08 (Estimated); Last update posted 2013-03-20 (Estimated); Status verified 2013-03

CONDITIONS: Osteopenia
Keywords: biomechanics; osteogenesis; osteoporosis; bone regeneration
MeSH Terms: conditions — Bone Diseases, Metabolic; Osteoporosis

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Low magnitude mechanical stimulation (Experimental): 10 minutes per day of low magnitude mechanical stimulation using a vibrating platform set at 0.3 g and 30 Hz
  Interventions: Device: Low magnitude mechanical stimulation
- 2 (Placebo Comparator): 10 minutes per day standing on sham low mechanical stimulation platform
  Interventions: Device: Sham low magnitude mechanical stimulation

INTERVENTIONS:
Device: Low magnitude mechanical stimulation — 10 minutes per day of low magnitude mechanical stimulation using a vibrating platform set at 0.3 g and 30 Hz
  Arms: Low magnitude mechanical stimulation
Device: Sham low magnitude mechanical stimulation — 10 minutes per day of low magnitude mechanical stimulation using a sham vibrating platform
  Arms: 2

SUMMARY:
The purpose of this study is to determine if daily low magnitude, high frequency whole body vibration can improve bone density in seniors.

DETAILED DESCRIPTION:
The treatment options for osteoporosis, a major health complication in the aged population, are limited to pharmacologic interventions, the majority of which are antiresorptive. Preliminary data demonstrate that high frequency, low magnitude mechanical stimulation (LMMS) can preserve bone mineral density (BMD) by preventing bone resorption due to disuse and aging, and can stimulate new bone formation.

To confirm and extend these observations, this study is a three-year, double-blind, randomized, placebo-controlled clinical trial of LMMS in 200 elderly women and men (60 years of age and older). A clinical center located in Boston, MA has recruited participants from multiple independent living facilities in close geographic proximity. Participants meeting the inclusion/exclusion criteria have been randomized to either brief daily exposure to LMMS on a vibrating platform or a placebo platform over a three year period. All participants receive 1000 mg of elemental calcium and 800 IU of vitamin D per day.

This study will provide new and important information about the role of low magnitude high frequency mechanical stimulation on the skeleton.

ELIGIBILITY:
Inclusion Criteria:

* Men and women 60 years and over of all ethnic groups
* Weight less than 250 pounds
* Absence of terminal cancer or other illness necessitating hospice level services
* Capable of following the protocol and of understanding and providing informed consent
* Scoring less than 12 on the Short Blessed Test

Exclusion Criteria:

* Immobilization of the axial or lower appendicular skeleton within the last year
* Nonambulatory (ambulation with an assistive device will be permitted)
* Malignancy other than cured thyroid cancer or skin cancer
* Hip replacement or internal fixation, total knee replacement, or lower limb fracture within the past year, or bilateral hip replacement
* Medications: glucocorticoids, suppressive doses of thyroid hormone as determined by screening TSH, anticonvulsant drugs (phenytoin, phenobarbital, carbamazepine), estrogen/testosterone replacement, selective estrogen receptor modulators (SERMs), PTH, or bisphosphonates more than 1 month in past year, calcitonin therapy within the preceding month, fluoride therapy at any time
* Paget's disease of bone, rheumatoid arthritis or other connective tissue disorders requiring systemic treatment with disease modifying drugs, or a history of Cushing's syndrome
* Fragility fracture within the past five years unless pharmacologic therapy not to be prescribed

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 174 (Actual)
Dates: Start 2007-02; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Changes in volumetric trabecular BMD of the spine and hip by quantitative computed tomography (CT scan) | 2 - 3 years

SECONDARY OUTCOMES:
Changes in biochemical markers of bone formation (Procollagen type 1 N-terminal peptide and Bone Specific Alkaline Phosphatase) and resorption (C-terminal Telopeptide of type I collagen) | 2 - 3 years
Changes in postural stability | 2 - 3 years
  Postural stability measured as quiet stance with eyes open for 4 minutes on a Kistler force platform
Changes in isometric leg extension strength | 2 - 3 years
  Isometric knee extension strength of the right leg measured with a handheld dynamometer
Change in hip muscle area and density | 2 - 3 years
  Muscle area and density surrounding the hips measured by quantitative computed tomography

CONTACTS AND LOCATIONS:
Overall Officials: Douglas P. Kiel, MD, MPH, Principal Investigator — Institute for Aging Research, Hebrew SeniorLife; Marian T. Hannan, DSc, MPH, Principal Investigator — Institute for Aging Research, Hebrew SeniorLife
Locations (1):
- Hebrew SeniorLife, Institute for Aging Research, Boston, Massachusetts, United States

REFERENCES:
- [Background] Ward K, Alsop C, Caulton J, Rubin C, Adams J, Mughal Z. Low magnitude mechanical loading is osteogenic in children with disabling conditions. J Bone Miner Res. 2004 Mar;19(3):360-9. doi: 10.1359/JBMR.040129. Epub 2004 Jan 27. PMID 15040823
- [Background] Rubin C, Recker R, Cullen D, Ryaby J, McCabe J, McLeod K. Prevention of postmenopausal bone loss by a low-magnitude, high-frequency mechanical stimuli: a clinical trial assessing compliance, efficacy, and safety. J Bone Miner Res. 2004 Mar;19(3):343-51. doi: 10.1359/JBMR.0301251. Epub 2003 Dec 22. PMID 15040821
- [Background] Gilsanz V, Wren TA, Sanchez M, Dorey F, Judex S, Rubin C. Low-level, high-frequency mechanical signals enhance musculoskeletal development of young women with low BMD. J Bone Miner Res. 2006 Sep;21(9):1464-74. doi: 10.1359/jbmr.060612. PMID 16939405
- [Background] Kiel DP, Hannan MT, Barton BA, Bouxsein ML, Lang TF, Brown KM, Shane E, Magaziner J, Zimmerman S, Rubin CT. Insights from the conduct of a device trial in older persons: low magnitude mechanical stimulation for musculoskeletal health. Clin Trials. 2010 Aug;7(4):354-67. doi: 10.1177/1740774510371014. Epub 2010 Jun 22. PMID 20571129
- [Derived] Muir JW, Kiel DP, Hannan M, Magaziner J, Rubin CT. Dynamic parameters of balance which correlate to elderly persons with a history of falls. PLoS One. 2013 Aug 5;8(8):e70566. doi: 10.1371/journal.pone.0070566. Print 2013. PMID 23940592
- [Derived] Jeffrey BA, Hannan MT, Quinn EK, Zimmerman S, Barton BA, Rubin CT, Kiel DP. Self-reported adherence with the use of a device in a clinical trial as validated by electronic monitors: the VIBES study. BMC Med Res Methodol. 2012 Nov 14;12:171. doi: 10.1186/1471-2288-12-171. PMID 23150931